CLINICAL TRIAL: NCT05118841
Title: A Phase 1, Open-Label, First in Human, Dose Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of ZX-4081 in Patients With Advanced Solid Tumors
Brief Title: Dose-Escalation and Dose-Expansion Study of ZX-4081 in Patients With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing Zenshine Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ZX-4081
Record Dates: First submitted 2021-10-18; First posted 2021-11-12 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- ZX-4081 Dose Level 1 (Experimental): Starting dose (SD) of ZX-4081 administered orally twice daily (BID) in a 28-day cycle
  Interventions: Drug: ZX-4081
- ZX-4081 Dose Level 2 (Experimental): 2-times the SD of ZX-4081 administered orally BID in a 28-day cycle
  Interventions: Drug: ZX-4081
- ZX-4081 Dose Level 3 (Experimental): 4-times the SD of ZX-4081 administered orally BID in a 28-day cycle
  Interventions: Drug: ZX-4081
- ZX-4081 Dose Level 4 (Experimental): 6-times the SD of ZX-4081 administered orally BID in a 28-day cycle
  Interventions: Drug: ZX-4081
- ZX-4081 Dose Level 5 (Experimental): 8-times the SD of ZX-4081 administered orally BID in a 28-day cycle
  Interventions: Drug: ZX-4081
- ZX-4081 Dose Level 6 (Experimental): 10-times the SD of ZX-4081 administered orally BID in a 28-day cycle
  Interventions: Drug: ZX-4081
- ZX-4081 Expansion Dose Level (Experimental): Recommended Phase 2 Dose (RP2D) (to be determined) of ZX-4081 administered orally BID in a 28-day cycle
  Interventions: Drug: ZX-4081

INTERVENTIONS:
Drug: ZX-4081 — Twice daily (BID), oral dosing of ZX-4081 at the assigned dose level in a 28-day cycle

SUMMARY:
A Phase 1, first-in-human, open-label, multicenter, dose escalation and dose expansion study to investigate the safety, tolerability, PK, pharmacodynamics, and preliminary antitumor activity of ZX-4081 administered orally (PO) twice daily (BID) in 28-day cycles in patients with Advanced Solid Tumors.

ELIGIBILITY:
Inclusion Criteria:

1. Metastatic or locally advanced solid tumor malignancies (breast cancer, urothelial cancer, ovarian cancer, melanoma, NSCLC, renal cell carcinoma, squamous cell cancer of the head and neck, colorectal cancer, and hepatocellular carcinoma) that has progressed on, is refractory to, intolerant to, or for which there is no curative standard of care therapy.
2. Measurable disease with at least 1 lesion amenable to response assessment per RECIST 1.1.
3. Demonstrate adequate organ function. All screening laboratories should be performed within 14 days of treatment initiation.
4. Has a performance status of 0-2 on the ECOG Performance Scale.
5. Life expectancy >12 weeks at baseline.
6. Women of childbearing potential must have negative serum or urine pregnancy test within 72 hours prior to receiving the first study drug administration. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

   Women of childbearing potential must be willing to use an adequate method of contraception from 30 days prior to the first study drug administration and 120 days following last day study drug administration.
7. Male patients of childbearing potential must be surgically sterile, or must agree to use adequate method of contraception during the study and at least 120 days following the last day of study drug administration.
8. Age ≥18 years at screening.
9. Able and willing to provide written informed consent and to follow study instructions.

Exclusion Criteria:

1. Patient has disease that is suitable for therapy administered with curative intent.
2. Untreated or uncontrolled central nervous system (CNS) involvement.
3. Any concurrent or recent use (within 28 days or 5 half-lives, whichever is longer) of chemotherapy, immunotherapy, or biologic or hormonal therapy for cancer treatment.
4. Unresolved toxicities from prior therapy, defined as having not resolved to NCI CTCAE v5.0 Grade 0 or 1, with exception of alopecia and vitiligo.
5. Systemic corticosteroids at doses exceeding 10 mg/day prednisone or equivalent.
6. Patient has an active infection requiring systemic therapy.
7. Patients who have known active HIV, Hepatitis or active COVID-19 infection. (Patients who have been vaccinated against Hepatitis B and who are positive only for the Hepatitis B surface antibody are permitted to participate in the study). Patients who are positive for hepatitis B or C virus must be tested for and have an undetectable viral load.
8. Patients with unstable/inadequate cardiac function:

   1. New York Heart Association Class 3 or 4 congestive heart failure,
   2. Uncontrolled hypertension,
   3. Acute coronary syndrome within 6 months,
   4. Clinical important cardiac arrhythmia,
   5. A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >470 milliseconds (ms) (CTCAE grade 1) using Fredericia's QT correction formula.
9. A history of additional risk factors for Torsades de Pointes(TdP) (e.g., heart failure, hypokalemia, family history of Long QT Syndrome).
10. The use of concomitant medications that prolong the QT/QTc interval.
11. Concomitant use or recent use (at least 2 weeks before the start of ZX-4081 treatment) of drugs that are known to be strong CYP3A4/5 inhibitors and CYP3A4/5 inducers (See 5.4.2 for a list of study medications not allowed during this study).
12. Concomitant use of drugs that are sensitive substrates with narrow therapeutic index for one of the following: CYP2C9, CYP2C19, CYP2C8, CYP2D6 and CYP3A4 (See 5.4.2 for a list of study medications not allowed during this study).
13. Concomitant use of drugs that are sensitive substrates with narrow therapeutic index for one of the following transporters: P-glycoprotein (P-gp) and Breast Cancer resistance Protein (BCRP).
14. Recent use a proton pump inhibitor (within 4 days prior to the start ZX-4081 treatment) or a histamine H2 blocker (within 2 days prior to the start of ZX-4081 treatment).
15. Uncontrolled concurrent illness.
16. Patient has concurrent active malignancy other than nonmelanoma skin cancer, carcinoma in situ of the cervix, or superficial bladder cancer who has undergone potentially curative therapy with no evidence of disease. Patients with other previous malignancies are eligible if disease-free for >2 years.
17. Participation in another clinical trial of an investigational agent within 30 days of screening.
18. Patient has known psychiatric, substance abuse or other disorders that would interfere with cooperation with the requirements of the trial, in the opinion of the investigator.
19. Patients who are pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 30 days after the last dose of trial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-01-03 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Determine the recommended Phase 2 dose (RP2D) of ZX-4081 | At the end of Cycle 1 (each cycle is 28 days)
  To assess number of patients experiencing dose-limiting toxicities (DLTs) in the dose escalation phase
Safety and tolerability of ZX-4081 | From first dose of ZX-4081 through 28 days after the last ZX-4081 treatment (up to 2 years); each cycle is 28 days
  To examine the incidence of clinical and laboratory adverse events after multiple doses of ZX-4081 in the dose escalation and dose expansion phases

SECONDARY OUTCOMES:
Peak Plasma Concentration of ZX-4081 | Days 1, 8, and 15 of Cycle 1 (each cycle is 28 days)
  To evaluate the maximum observed concentration (Cmax) after single and repeated oral, twice daily (BID) doses of ZX-4081
Area under the plasma concentration of ZX-4081 | Days 1, 8, and 15 of Cycle 1 (each cycle is 28 days)
  To evaluate the area under the curve (AUC) plasma-concentration after single and repeated oral, BID doses of ZX-4081
Half-life of ZX-4081 | Days 1, 8, and 15 of Cycle 1 (each cycle is 28 days)
  To evaluate the half-life of ZX-4081 after single and repeated oral, BID doses of ZX-4081
Objective response rate (ORR) | Up to 2 years
  To evaluate the objective response rate (ORR) as determined by the specific disease response criteria
Duration of Response (DOR) | Up to 2 years
  To examine the duration of response (DoR), defined as time from the date of first documentation of response to the date of the first documentation of progressive disease (PD), or death due to any cause
Progression Free Survival (PFS) | Up to 2 years
  To examine the the progression free survival (PFS), defined as time from the date of first dose of study treatment to the first date of documentation of PD, or death due to any cause
Overall Survival (OS) | Up to 2 years
  To examine the overall survival (OS), defined as time from the date of first dose of study treatment to death due to any cause
Peripheral myeloid-derived suppressor cell (MDSC) proportion in the blood | Cycle 1 Day1 , Cycle 2 Day 1, and Cycle 3 Day 1 (each cycle is 28 days)
  To assess the changes of peripheral MDSC proportion in the blood after single and repeated oral, BID doses of ZX-4081
T cell composition and activation status | Cycle 1 Day1 , Cycle 2 Day 1, and Cycle 3 Day 1 (each cycle is 28 days)
  To assess the impact on T cell profiles after repeated oral, BID doses of ZX-4081

CONTACTS AND LOCATIONS:
Locations (1):
- Carolina BioOncology, Huntersville, North Carolina, United States